CLINICAL TRIAL: NCT04901455
Title: Nasal Mucosal Immune Responses to Live Attenuated Influenza Virus (LAIV) in Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Phenotypes
Brief Title: Responses to Live Attenuated Influenza Virus (LAIV) in Chronic Obstructive Pulmonary Disease (COPD)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-0254; 1R01HL150081-01A1 (NIH)
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — FluMist

STUDY DESIGN:
Intervention Model Description: This study is an early Phase 1, single-center, parallel-group unmasked exposure study of nasal immune responses after controlled exposure to LAIV.
Masking Description: This is an open label exposure study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- COPD Frequent Exacerbators (Experimental): Individuals with two or more episodes of worsening in COPD symptoms requiring treatment with antibiotics and/or steroids in the prior 12 months
  Interventions: Biological: LAIV
- COPD Infrequent Exacerbators (Experimental): Individuals with less than two episodes of worsening in COPD symptoms requiring treatment with antibiotics and/or steroids in the prior 12 months
  Interventions: Biological: LAIV
- Healthy Control (Experimental): Individuals with spirometry-confirmed normal lung function and no asthma history
  Interventions: Biological: LAIV

INTERVENTIONS:
Biological: LAIV — Standard dose of LAIV administered by a licensed health care providers.
  Other Names: FluMist

SUMMARY:
This study will determine the functional status of the nasal immune environment with LAIV exposure in COPD persons with frequent exacerbations (defined as individuals with two or more episodes of worsening in COPD symptoms requiring treatment with antibiotics and/or steroids in the prior 12 months) and COPD persons without frequent exacerbations to determine acute exacerbation of COPD (AECOPD)-associated dysfunction in a) cytokines and immune effector cells of the nasal mucosa and b) viral replication. The investigators hypothesize that: 1) COPD frequent exacerbators, compared to COPD infrequent exacerbators, will demonstrate altered mucosal immune responses to LAIV exposure, and 2) COPD frequent exacerbators, compared to COPD infrequent exacerbators, will demonstrate increased markers of influenza viral replication after LAIV exposure.

DETAILED DESCRIPTION:
This study is an early Phase 1, single-center, single-group unmasked exposure study of nasal immune responses after controlled exposure to LAIV. This trial will test the differences in the nasal immune responses to the nasal flu vaccine in two diseased groups of individuals along with healthy controls: COPD persons with frequent exacerbations (defined as individuals with two or more episodes of worsening in COPD symptoms requiring treatment with antibiotics and/or steroids in the prior 12 months) and COPD persons without frequent exacerbations (defined as individuals with less than two episodes of worsening in COPD symptoms requiring treatment with antibiotics and/or steroids in the prior 12 months). A healthy control cohort will also be recruited, defined as individuals with spirometry-confirmed normal lung function and no asthma history. A total of 15 COPD frequent exacerbators, 15 infrequent exacerbators and 10 healthy controls will be enrolled for this trial. Investigators will balance the sex of participant as closely as possible to 50% male and 50% female.

At screening visit, after obtaining informed consent and authorization to obtain medical records, all potential individuals will be screened for specific inclusion and exclusion criteria to ensure suitability and safety to receive the influenza nasal vaccine. A baseline assessment will be done including reviewing medical history and verifying eligibility, a physical exam by a study investigator, spirometry testing before and after bronchodilator, laboratory testing to screen for immunocompromised state [Human Immunodeficiency Virus (HIV) antibody testing, compete blood count (CBC) with differential], an assessment of symptoms, and pregnancy testing if pre-menopausal. Women who are pregnant, nursing, or women who are currently trying to become pregnant are not eligible for this study.

Participants who meet eligibility after screening will be brought back for an enrollment visit where they will undergo a baseline assessment of their nasal inflammatory state. This includes sampling of the nose in three different ways. First, investigators will gently place a small strip of absorbent paper inside the lower part of the nose, and a nose clip will be applied for two minutes (ELF collection). Next, investigators will wash the inside of the nose with a small amount of sterile salt water to collect samples (NLF collection). Finally, investigators will take a small plastic device and gently scrape the inside of the nose to collect nasal cells (scraping collection). Investigators will also collect blood samples for inflammatory phenotyping.

Within two weeks of enrollment visit, all enrolled individuals will receive the nasal influenza vaccine (there is no placebo component to the study). On days one, two, three, and seven after vaccine administration, participants will return to the study site to undergo nasal sampling including the nasal paper strip and washing, as well as blood collection. On Day 3, a nasal scraping will also be obtained. On Day 21 (optional visit), investigators will obtain nasal washing and blood collection. Investigators will collect patient reported outcomes using a validated influenza severity score to assess for unbiased correlations with biological measures.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual in the COPD group must meet all of the following criteria:

* Age>40 years old
* Physician diagnosis of COPD confirmed by post-bronchodilator testing (defined as forced expiratory volume in one second (FEV1)/forced vital capacity (FVC)< lower limit of normal and FEV1/FVC<0.70) and FEV1>30% predicted based on spirometry testing available in the prior year or completed at screening (if no historical testing available)
* Free of acute exacerbation of COPD for prior four weeks at time of recruitment
* Resting oxygen saturation >94 percent
* Blood pressure systolic values between 90-160 mm Hg and diastolic between 55-90 mm Hg
* No nasal symptoms based on questionnaire
* Willingness and ability to participate in study procedures
* Completion of informed consent

In order to be eligible to participate in this study, an individual in the healthy control group must meet all of the following criteria:

* Age>40 years old
* Spirometry testing showing normal lung function (defined as pre and post--bronchodilator FEV1/FVC>=lower limit of normal and FEV1>80 percent predicted) based on spirometry testing available in the prior year or completed at screening (if no historical testing available)
* Resting oxygen saturation >94 percent
* Blood pressure systolic values between 90-160 mm Hg and diastolic between 55-90 mm Hg
* No nasal symptoms based on questionnaire
* Willingness and ability to participate in study procedures
* Completion of informed consent

Exclusion Criteria:

* Inability or unwillingness to consent
* Active tobacco or e-cigarette use (within last six months)
* Active diagnosis of asthma
* Any regular suppressive antibiotics (i.e., azithromycin)
* Daily oral prednisone use
* Any supplemental oxygen use beyond nocturnal oxygen therapy
* Use of intranasal corticosteroids in the 30 days prior to screening visit
* Chronic illness associated with immunosuppression (i.e., HIV, malignancy)
* History of documented or self-reported positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection requiring hospitalization
* Receipt of SARS-CoV-2 vaccine within 14 days prior to study screening visit or plan to receive SARS-CoV-2 vaccine from screening visit to 14 days after completion of all study procedures
* History of epistaxis, prior nasal surgery or anatomical abnormalities
* Current use of blood thinner beyond full dose aspirin [e.g., warfarin (coumadin), clopidogrel (Plavix), dabigatran (Pradaxa), rivaroxaban (Xarelto), apixaban (Eliquis)]
* Self-reported history of easy bruising or bleeding gums
* Serological evidence of HIV infection at screening (Positive HIV antibody test)
* Relative leukopenia (WBC<4000), neutropenia (Absolute neutrophil count<2000) or lymphopenia (absolute lymphocyte count<1500) on screening CBC
* Respiratory infection (cough, sore throat, sinusitis, fever) within prior 4 weeks
* Active wheezing at day 0 visit
* Pregnancy or nursing or women who are currently trying to become pregnant. (All female subjects, except those who have had a hysterectomy with oophorectomy, will undergo urine pregnancy testing on the morning of the screening visit and again on the on Day 0 at the time of arrival to the lab and prior to LAIV administration. A positive pregnancy test will exclude the subject)
* Use of chronic immunosuppression in the 30 days prior to screening visit
* History of hypersensitivity, especially anaphylactic reactions, to egg proteins, gentamicin, gelatin, or arginine, or with a reaction to previous influenza vaccination at a severity level precluding the subject's participation as judged by the study physician
* History of Guillain-Barre syndrome
* Subjects who will be unable to avoid contact with immunocompromised individuals for 3 weeks after receiving LAIV vaccine
* Receipt of the LAIV during the current or prior flu vaccine season
* Physician diagnosed influenza, a positive test for influenza or suspicion of influenza illness in the 18 months prior to enrollment. Suspicion of influenza will be based on the CDC's influenza-like illness case definition ("fever>100 °F AND cough/sore throat in the absence of a known cause other than influenza. Temperature can be measured in the office or at the home")
* Any condition that, in the opinion of the study investigator, would compromise the subject's ability to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Difference in mucosal immune response between COPD frequent exacerbators and COPD infrequent exacerbators | Baseline, Day 3
  Epithelial lining fluid interferon-gamma (INF-ɣ) area under the curve (AUC) from day 0 (baseline) to day 3 (pg/mL x days)

SECONDARY OUTCOMES:
Difference in viral clearance between COPD frequent exacerbators and COPD infrequent exacerbators | Baseline, Day 3
  Nasal scrape influenza gene expression AUC from day 0 (baseline) to day 3

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Drummond, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Eastowne Medical Office Building, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months following publication through 36 months after publication
Access Criteria: Proposing investigator has IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.